CLINICAL TRIAL: NCT01720836
Title: Study of the Immunogenicity of the MUC1 Peptide - Poly-ICLC (Polyinosinic-polycytidylic Acid Stabilized With Polylysine and Carboxymethylcellulose) OR HILTONOL™ Adjuvant Vaccine in Patients With Localized and Locally Advanced Non-Small Cell Lung Cancer
Brief Title: Study of the Immune Response of MUC1 (Mucin1) Peptide Vaccine for Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Olivera Finn (Other)
Responsible Party: Sponsor-Investigator, Olivera Finn, Professor of Immunology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-094; 902168 (Other Grant/Funding Number: V Foundation)
Record Dates: First submitted 2012-10-31; First posted 2012-11-02 (Estimated); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (3):
- Stage IA or I/II NSCLC or neuroendocrine carcinoid tumor (Experimental): Resection or radiotherapy without adjuvant chemotherapy followed by 3 cycles of vaccine + PolyICLC.
  Interventions: Biological: Vaccine + PolyICLC
- Stage IB/II/IIIA (Experimental): Resection and adjuvant chemotherapy followed by 3 cycles of vaccine + PolyICLC.
  Interventions: Biological: Vaccine + PolyICLC
- Stage IIIA or IIIB (Experimental): Concomitant chemo-irradiation followed by 3 cycles of vaccine + PolyICLC.
  Interventions: Biological: Vaccine + PolyICLC

INTERVENTIONS:
Biological: Vaccine + PolyICLC — The vaccine will consist of 100 micrograms of MUC1 100mer peptide dissolved in 50 micro-liters of sterile saline, admixed with 500 micrograms of Hiltonol® in 250 microliters volume, for a total injection volume of 300 microliters.

SUMMARY:
All subjects will receive the vaccine subcutaneously every 3 weeks x 3 with optional yearly booster vaccines up to and including 5 years post last vaccine for those patients who are confirmed responders to the vaccine . The rationale for using Poly-ICLC as an adjuvant are two ongoing trials at University of Pittsburgh Cancer Institute (UPCI) of the MUC1 100mer peptide vaccine - one as a therapeutic vaccine in subjects with metastatic castrate resistant prostate cancer and the other in subjects with advanced colonic adenomas at risk for developing colon cancer. The same formulation, MUC1 100mer peptide admixed with Poly-ICLC, is used in both trials. There has been no toxicity observed and the vaccine is highly immunogenic in early disease. In the proposed NSCLC trial the anti-MUC1 immune response will be thoroughly characterized.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC) or neuroendocrine carcinoid tumor
* All subjects must have one of the following stages: Stage IA(T1NO); IB (T2NO), II & IIIA (N2 negative); IIIA (N2+), IIIB (N3+)
* Patients must have stable disease at the time of enrollment
* Women and men at least 18 years of age
* ECOG performance status 0-1(Appendix A)
* Subjects must be within 4 to 24 weeks of standard of care treatment for their particular stage of disease
* Subjects must have acceptable organ and marrow function as defined below:

  * Leukocytes > 3,000/µL
  * Absolute Neutrophils > 1,500/µL
  * Hemoglobin > 10 g/dL
  * Platelets > 100,000/µL
  * Total Bilirubin within normal institutional limits
  * Creatinine within normal institutional limits OR
  * Creatinine clearance > 60 mL/min/1.73 m2 for subjects with above normal AST and ALT with alkaline phosphatase within < 1.5 times upper limit of normal
* The effects of a MUC1vaccine on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, men and women of childbearing potential must be willing to use effective contraception (hormonal barrier method of birth control; abstinence) while on study treatment and for at least 3 months thereafter. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria:

* Subjects may not be receiving any other investigational agents

  - No history of prior malignancy, except for non-melanoma skin cancer
* Any positive ANA titer above 1:160, even in an asymptomatic individual. Note:

Weakly positive ANA defined as ANA titers up to 1:160 maximum (≤ 1:160) will be acceptable in an asymptomatic individual who is otherwise eligible for the study.

* Known Hepatitis B on immunomodulators (i.e. interferon)
* Known Hepatitis C on immunomodulators (i.e. interferon)
* No prior vaccine therapy
* Patients may not be receiving any steroids or other anti-immune therapy at the time of registration.
* Subjects must not be more than 24 weeks from standard of care treatment for their particular stage of disease
* Subjects must not have post-obstructive pneumonia or other serious infection at the time of registration or other serious underlying medical condition that would impair the ability of the subjects to receive protocol treatment
* Prior resection of lung cancer is allowed, if at least five years have elapsed between previous resection and registration
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study. Women of childbearing potential must have a negative pregnancy test
* Subjects with immune deficiency are not expected to respond to the vaccine. Therefore, known HIV-positive patients are excluded from the study
* Subjects with a history of known autoimmune disease are excluded from this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-11; Primary Completion 2027-10 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Immunologic response | 2 years
  Immunologic response will be measured by increases in anti MUC1 antibody titers post vaccination at different stages of disease: localized (Stage I, II) or locally advanced (Stage III) non-small cell lung cancer and neuroendocrine carcinoid tumors.

SECONDARY OUTCOMES:
Anti-MUC1 immunity | 2 years
  To assess spontaneous anti- MUC1 immunity in response to cancer prior to administration of the MUC1 vaccine
Association between baseline MUC1 immunity and vaccine | 2 years
  To assess the association between baseline MUC1 immunity and vaccine - induced increases in anti MUC1 antibodies
Immunocompetence versus immunosuppression | 2 years
  To characterize the change in the balance between immunocompetence (response of T cells to polyclonal stimulation) versus immunosuppression at different stages of disease {check for increased numbers of regulatory T cells (Treg) and Myeloid-Derived Suppressor Cells (MDSC)}
MUC1 associated safety | 2 years
  To monitor adverse events associated with the study agents
survival | 2 years
  To monitor for progression free survival
survival | 2 years
  To monitor for progression of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Arjun Pennathur, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States